CLINICAL TRIAL: NCT01473264
Title: Safety and Tolerability of Recombinant Human Clara Cell 10kDa Protein (rhCC10) Delivered Intratracheally to Premature Neonates With Respiratory Distress Syndrome
Brief Title: Safety, Pk and Anti-inflammatory Effects of CC10 Protein in Premature Infants With Respiratory Distress Syndrome (RDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clarassance, Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CC10-2000-001; 9R44HL066965-02 (NIH)
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Respiratory Distress Syndrome in Premature Infant; Bronchopulmonary Dysplasia
Keywords: CC10; BPD; Bronchopulmonary dysplasia; premature infants; neonates; pulmonary inflammation; lung function; RDS
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth; Pneumonia | interventions — Uteroglobin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator)
  Interventions: Drug: placebo
- High dose rhCC10 (Experimental): 5 mg/kg study drug (rhCC10)
  Interventions: Drug: recombinant human CC10 (rhCC10)
- Low Dose rhCC10 (Experimental): 1.5 mg/kg study drug (rhCC10)
  Interventions: Drug: recombinant human CC10 (rhCC10)

INTERVENTIONS:
Drug: recombinant human CC10 (rhCC10) — 5 mg/kg rhCC10, single dose delivered intratracheally (IT). Treatment was delivered within four hours after surfactant treatment. Dose was delivered IT in two (2) equal aliquots via a premeasured feeding tube placed in the distal third of the endotracheal tube with the patient in the right and then left lateral decubitus position and 30 degrees of Trendelenburg.
  Other Names: rhCC10; CC10; uteroglobin; Clara cell secretory protein; Clara cell 10 kDa protein
  Arms: High dose rhCC10
Drug: recombinant human CC10 (rhCC10) — 1.5 mg/kg rhCC10, single dose delivered intratracheally (IT). Treatment was delivered within four hours after surfactant treatment. Dose was delivered IT in two (2) equal aliquots via a premeasured feeding tube placed in the distal third of the endotracheal tube with the patient in the right and then left lateral decubitus position and 30 degrees of Trendelenburg
  Other Names: rhCC10; CC10; uteroglobin; Clara cell secretory protein; Clara cell 10 kDa protein
  Arms: Low Dose rhCC10
Drug: placebo — Half normal saline solution; single dose delivered intratracheally (IT). Treatment was delivered within four hours after surfactant treatment. Dose was delivered IT in two (2) equal aliquots via a premeasured feeding tube placed in the distal third of the endotracheal tube with the patient in the right and then left lateral decubitus position and 30 degrees of Trendelenburg.
  Arms: Control

SUMMARY:
Bronchopulmonary Dysplasia (BPD) is a multi-factorial disease process that is the end result of an immature, surfactant deficient lung that has been exposed to hyperoxia, mechanical ventilation and infection. These conditions initiate an inflammatory response characterized by elevated inflammatory cell infiltrates and proinflammatory cytokines that lead to the development of significant acute and chronic lung injury.

The study drug, rhCC10, is a recombinant version of natural human CC10 protein. Native CC10 is produced primarily by non-ciliated respiratory epithelial cells, called Clara cells and is the most abundant protein in the mucosal fluids in normal healthy lungs.

The purpose of this study was to evaluate the pharmacokinetics, safety, tolerability and anti-inflammatory effects of a single intratracheal (IT) dose of rhCC10 to intubated premature infants receiving positive pressure ventilation for treatment of respiratory distress syndrome (RDS) to prevent long term respiratory complications referred to as bronchopulmonary dysplasia, and, more recently, as chronic respiratory morbidity (CRM; asthma, cough, wheezing, multiple respiratory infections).

CC10 regulates inflammatory responses and protects the structural integrity of pulmonary tissue while preserving pulmonary mechanical function during various insults (eg. viral infection, bacterial endotoxin, ozone, allergens, hyperoxia). Together these properties suggest that administration of rhCC10 may help to facilitate development of normal airway epithelia and prevent the inflammation that leads to CRM in these infants.

ELIGIBILITY:
Inclusion Criteria:

Newborn infants were considered for the study if the following criteria were met:

* Age < 24 hours;
* Birthweight between 700 and 1,300 grams;
* Gestational age greater than or equal to 24 weeks;
* Diagnosis of neonatal RDS based on clinical and radiographic criteria;
* Requiring intubation and mechanical ventilation for treatment of RDS;
* Received at least one dose of surfactant 100 mg/kg (Survanta; Ross Laboratories);
* Written informed consent from the infant's parent or legal guardian prior to enrollment of the patient and agrees to all study-related procedures and evaluations, including those required after hospital discharge.

Exclusion Criteria:

• Major congenital abnormalities (chromosomal, genetic, cardiac, pulmonary, or renal);

Ages: 24 Weeks to 29 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2000-01; Primary Completion 2002-06 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Number and type of adverse events | Adverse events were monitored through 36 wks post-menstrual age (PMA) or hospital discharge
  All adverse events were monitored according to the NCI Common Toxicity Criteria. In addition, adverse events specific to, or likely to occur in, premature infants were also monitored, including apnea/bradycardia, sepsis (culture-confirmed), patent ductus arteriosus, retinopathy of prematurity, intraventricular hemorrhage, periventricular leukomalacia, and necrotizing enterocolitis (NEC).

SECONDARY OUTCOMES:
Assessment of pulmonary inflammatory markers | Days 0-7
  Total cell and neutophil counts were performed on TAF fluids. In addition, a panel of cytokines were measured in TAF from patients at times 0, 1, and 2 days
Total number of days on mechanical ventilation | Through 36 wks postmenstrual age or discharge
Hospitalization at 36 weeks PMA | Through 36 wks postmenstrual age or discharge
Chronic Respiratory Morbidity | 6 & 12 months postmenstrual age
  Physical exams and Bayley neurological exams were performed at 12 months PMA. Data pertaining to respiratory outcomes were collected at 6 and 12 months PMA.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Davis, MD, Principal Investigator — Dept of pediatrics, Winthrop University Hospital, SUNY Stony Brook School of Medicine; Ira Gewolb, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - Christiana HealthCare Systems, Wilmington, Delaware
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Winthrop-University Hospital, SUNY Stony Brook School of Medicine, Mineola, New York

REFERENCES:
- [Result] Levine CR, Gewolb IH, Allen K, Welch RW, Melby JM, Pollack S, Shaffer T, Pilon AL, Davis JM. The safety, pharmacokinetics, and anti-inflammatory effects of intratracheal recombinant human Clara cell protein in premature infants with respiratory distress syndrome. Pediatr Res. 2005 Jul;58(1):15-21. doi: 10.1203/01.PDR.0000156371.89952.35. Epub 2005 Mar 17. PMID 15774846